CLINICAL TRIAL: NCT02822560
Title: Comparative Clinical and Economic Analysis of Percutaneous vs. Open Access for Endovascular Aortic Repair - a Prospective, Randomised Trial.
Brief Title: Economic Comparison of Percutaneous (pEVAR) vs. Open Access in EVAR.
Acronym: EVAccess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Responsible Party: Principal Investigator, Miriam Uhlmann, M.D., Wilhelminenspital Vienna
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-014-0216
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Aortic Aneurysm
Keywords: Endovascular Aortic Repair (EVAR); percutaneous EVAR (pEVAR); cost analysis; procedure time
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- pEVAR (Active Comparator): percutaneous femoral access using a suture-mediated closure system
  Interventions: Device: pEVAR
- open femoral access (Active Comparator): cutdown to femoral artery and surgical closure
  Interventions: Procedure: open femoral access

INTERVENTIONS:
Device: pEVAR — percutaneous femoral access using a suture-mediated closure device
  Arms: pEVAR
Procedure: open femoral access — cutdown to femoral artery and surgical closure
  Arms: open femoral access

SUMMARY:
The present clinical trial is performed in the field of vascular surgery. The aim of the study is the economical and clinical comparison of two different access ways to the femoral artery with intention of endovascular repair of aortic aneurysm. The usual access is a surgical cutdown to the femoral artery and is compared to a percutaneous access which is closed via a suture mediated device (Perclose ProGlide, Abbott).

DETAILED DESCRIPTION:
Introduction:

Endovascular repair of aortic aneurysms (EVAR) is a routine procedure in vascular surgery and associated with less perioperative complications compared to open aortic repair. Continuous improvement of endovascular techniques is crucial for sufficient patient care, especially in elderly with serious comorbidities. Percutaneous access (pEVAR) to the femoral artery is associated with less wound complications when performed in suitable patients. Prospective data about economic feasibility and exact duration of the technique itself compared to the open access during the surgery are missing.

Methods and data collection:

The primary endpoints of this prospective randomised single center trial are cost and time differences of open vs. percutaneous access. Each Patient enrolled in the study will receive percutaneous on one side and surgical access on the other side of the groin for femoral artery access.

The punction site will be closed using the Perclose ProGlide Suture-Mediated Closure System manufactured by Abbott Vascular. This device works through stiff wire guided delivering of a monofilament suture to the femoral artery punction site. After finishing endovascular procedures for aneurysm repair, the thereby laid sutures are tightened to achieve hemostasis. This system is suitable for sheath sizes up to 21 F (.28 inch).

Open access on the other side is performed with a cutdown to the femoral artery and closure after finished procedure, with a polypropylene suture.

Patients who undergo endovascular aortic repair at the Department of Vascular Surgery of Wilhelminenspital Vienna are recruited for the study after informed consent and fulfilled inclusion criteria. Included are men and women from the age of 18 - 90 years with any indication for endovascular aneurysm repair (thoracic, infrarenal aortic or iliac artery aneurysm, or combinations of these). Indication for aneurysm repair is not a part of this study and is set in accordance to international guidelines. Women in childbearing years could be included after detailed explanation of special risks for further pregnancy after EVAR and after proof of negative pregnancy test. Exclusion criteria are occlusive aortic disease, aneurysm of the femoral artery, diameter < 5mm or severe calcification, patients with keloided inguinal site, adipositas per magna or demented patients.

Due to a prior power analysis a optimum number of 50 cases was determined. Randomization is performed by lot (patients draw an envelope which contains either left or right side is done by pEVAR).

Data is collected preoperatively with a case report form (CRF) including detailed health information about the patient. During the surgery, femoral artery access and wound closure time is measured separately for each side (in minutes). Material costs are also documented separately for each side (in €). Postoperative data about wound healing and pain of each inguinal side are collected descriptive using the CRF. Data management and analysis is anonymous using random patient numbers on the forms.

Main targets of the study are cost and time difference of percutaneous and open access techniques. Possible difference in both groups will be analyzed using the Wilcoxon Signed Rank Test. Postoperative data will be evaluated descriptively.

In case of cost advantage of the percutaneous access, this study economically legitimates the use of suture mediated closure systems and therefore contributes to the establishment of minimally invasive endovascular aortic repair.

ELIGIBILITY:
Inclusion Criteria:

* Indication for endovascular aortic repair

Exclusion Criteria:

* femoral aneurysm, severe femoral artery calcification, keloided inguinal region, severe obesity, patients diagnosed with Alzheimer's disease or severe psychiatric diagnosis, patient's with occlusive aortic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Overall costs of each different access | During surgery
  Overall costs of each different access way including used material and duration of the procedure (shorter duration = less costs of running operation theatre).

SECONDARY OUTCOMES:
Access duration | During surgery
  Separately measured duration of each access way itself (from start until first sheath is applied and from removal of sheath until wound is closed). The duration of endovascular repair is not included.

OTHER OUTCOMES:
Wound complications | up to 10 days postoperative
  Descriptive analysis of wound healing and complications after open vs. percutaneous access in the same individual.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, PD, MD, Study Director — Wilhelminenspital Vienna
Locations (1):
- Wilhelminenspital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Patient characteristics (gender, age, body mass index, earlier operations, written wound documentation etc.), operation time, material and overall procedure costs.

REFERENCES:
- [Derived] Uhlmann ME, Walter C, Taher F, Plimon M, Falkensammer J, Assadian A. Successful percutaneous access for endovascular aneurysm repair is significantly cheaper than femoral cutdown in a prospective randomized trial. J Vasc Surg. 2018 Aug;68(2):384-391. doi: 10.1016/j.jvs.2017.12.052. Epub 2018 Mar 8. PMID 29526378